CLINICAL TRIAL: NCT07311239
Title: Radiographic and Clinical Evaluation of Three-Dimensional Delta Plate in Internal Fixation of Mandibular Sub-condylar Fractures.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Collaborators: Ahmed Maher Teaching Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1299
Record Dates: First submitted 2025-11-16; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2024-11

CONDITIONS: Mandible Fracture
Keywords: Open Reduction and Internal Fixation of unilateral sub condylar fractures of the mandible; sub condylar fractures; 3D Delta Plate
MeSH Terms: conditions — Mandibular Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 14 patients recruited to the previously mentioned departments (Experimental)
  Interventions: Device: Three Dimensional Delta Plate

INTERVENTIONS:
Device: Three Dimensional Delta Plate — A 3D titanium plate designed with the following measurments: 1 mm thick, 20 mm long, 14 mm wide at the base, 5 mm wide at the apex. It has 4 holes where 2.00 mm screws can fit in.

SUMMARY:
In this study, we intend to examine the efficacy of 3D delta plates through radiographic evaluation of anatomic reduction and vertical ramus height as the main outcome and clinical assessment of pain and range of mandibular movements as secondary outcomes.

This Single arm longtudinal study will include 14 cases of trauma having mandibular sub condylar fractures, in which open reduction and internal fixation are indicated.

After selecting patients according to the inclusion criteria, all patients will undergo open reduction and rigid fixation.

Fracture will be stabilized using 4 hole, 2.0 mm 3-D Delta titanium plates using pre-auricular or retromandibular incision.

Radiographic evaluation using Computed Topograhy (CT) scans will be carried on immediatly after the operation then 3 months post operatively.

While, Clinical assessment will be performed at the following intervals after the surgery( 1 week, 1 month, 3 months)

DETAILED DESCRIPTION:
The study was conducted on fourteen patients suffering from unilateral mandibular subcondylar fractures gathered from Ain Shams University Department of Oral and Maxillofacial Surgery, Ahmed Maher Teaching Hospital and El-Bank El-Ahly Hospital for Integrated Care.

The used 3D plate is made of titanium, it is 1 mm thick, 20 mm long with a base measuring 14 mm and an apex measuring 5 mm. It has 4 holes (2 at the base and 2 at the top), where 2,00 mm screws can fit in.

The aim of this study is to evaluate the versatility of the three-dimensional delta plate in reduction and fixation of unilateral sub-condylar fractures. The results will be analyzed by radiographic assessment of proper anatomical reduction and measurement of vertical ramus height. In addition to, clinical outcomes of pain with jaw movements and measurement of all mandibular movements range.

Criteria of patients' selection :

Inclusion Criteria:

1. Patients at or over 18 years.
2. Unilateral sub condylar fractures indicated for treatment by open reduction and plate fixation according to valiati [55].

Exclusion Criteria:

1. Bilateral sub condylar fractures
2. Pediatric patients.
3. Intracapsular fractures
4. Patients with Uncontrolled systematic conditions.

Sample Size Calculation:

The sample size was estimated based on research published by Manoj et al. study (2015) regarding fracture fixation by trapezoidal 3D plate in India, by fixing alpha at 0.05 (5%) and beta at 0.05(5%), the minimal sample size is 10 patients to be included. To avoid drop out the sample was increased to 14 patients -Hypothesis: Delta plate doesn't provide an added advantage over the other Osteosynthesis methods of Sub condylar fixation.

Outcomes:

Primary outcomes: 1-Anatomic Reduction 2-Posterior Facial Height Secondary outcomes: 1-Pain 2-Mandibular Movements.

* Primary assessment of the patient:

  1- History:

  a. Personal History: Personal information was recorded for each patient, including name, age, sex, contact number, address, occupation, and marital status.

  b. Past Medical and Dental History: Relevant medical and dental history was documented, with particular attention to conditions that could influence treatment planning or pose risks during general anesthesia.

  c. History of Injury: Details regarding the injury were obtained from each patient, including the date and time of occurrence, any loss of consciousness at or following the event, the mechanism of injury, and the presence of any associated injuries

  2. Clinical Examination:
  1. General Condition on Admission:

     Airway patency and hemostasis were first ensured. The neurological status was assessed at presentation and categorized as clear, confused, or disoriented.
  2. Extraoral Examination:

     * Inspection: focused on identifying edema, ecchymosis, and gross deformity in regions suggestive of fracture. Associated soft-tissue injuries were documented, and the external auditory meatus was examined for evidence of blood or cerebrospinal fluid leakage.
     * Palpation: was conducted systematically from the condylar region along the entire mandibular border to detect tenderness, discontinuity of contour, or irregularity. In cases with suspected condylar fracture, digital palpation with the little finger in the external auditory meatus was employed to evaluate condylar head movement during mandibular excursions. Limitation of motion, pain, and localized tenderness were recorded, and neurosensory deficit of the lower lip, if present, was noted.
  3. Intraoral Examination:

     • Inspection: Saliva was examined for blood admixture. The buccal and lingual sulci were inspected for mucosal laceration, ecchymosis, or sublingual hematoma. Dental alignment was assessed, and mobility of individual teeth was documented. The occlusal plane was evaluated for step deformities suggestive of underlying fracture, and occlusion was examined for derangement or premature contact. Functional assessment of mandibular movements was performed to detect deviation, restriction, or pain.

     • Palpation: Bilateral palpation of the buccal and lingual sulci was undertaken to identify tenderness or step deformity. Finally, gentle bimanual manipulation of the mandible across suspected fracture sites was performed to elicit abnormal mobility.

     3-Radiographic examination: Computed tomograms (multi slice C.Ts) with three dimensional reconstructed images were obtained for all the patients.

     Radiographic evaluation was undertaken with the following objectives:

     1. To localize and determine the number of radiolucent fracture lines, and to identify additional fractures involving the mandible and adjacent facial bones.

     2. To exclude the presence of pathological lesions or foreign bodies that could potentially interfere with treatment planning.

     3. To assess the position of the fractured condylar segment and classify the condylar fracture according to the system of Lindahl and Hollender (1977).

     Preoperative Records:
     1. Demographic Data:

        Patient identifiers including name, age, sex, occupation, time of injury, and etiology of trauma were documented.
     2. Radiographic Records:

        Multi slice computed tomography (CT) with three-dimensional reconstruction was obtained for classification of condylar fractures and detection of associated maxillofacial fractures.
     3. Clinical Records:

  <!-- -->

  1. Standardized occlusal (frontal, right and left views) were recorded.
  2. Maximum painless, non-assisted and assisted interincisal distance was measured to assess mouth opening.
  3. Temporomandibular joint (TMJ) examination was performed, documenting pain and tenderness 4. Anesthetic Evaluation: It includes medical and surgical history, physical examination, investigations, risk assessment, consent and pre-medications.

     5.Antibiotic prophylaxis: No association was found between SSI and antibiotic prophylaxis for 24 hours or less vs 72 hours or more after OMF surgery.

     Treatment Phase:

     All patients were managed under general anesthesia by open reduction and internal fixation (ORIF) for subcondylar fractures and associated mandibular or midfacial fractures.

     Surgical Procedure for Subcondylar Fracture:
     1. General anesthesia was administered via nasotracheal intubation.
     2. Arch bars or intermaxillary fixation (IMF) screws were applied preoperatively, and maxillomandibular fixation was established.
     3. A modified retromandibular incision was marked, In the modified retromandibular approach, the area in the middle of the buccal and marginal mandibular branch of the facial nerve is utilized for dissection, thereby ensuring the protection of the facial nerve and preventing additional morbidity. The resultant scar is inconspicuous and satisfactory to the patient as it is almost always concealed in the retromandibular shadow. [85]
     4. Local infiltration with adrenaline (1:100,000) was administered along the incision line for hemostasis.
     5. After sterile preparation and draping, the skin was incised. Subcutaneous dissection was performed superficial to the superficial muscular aponeurotic system (SMAS) in an anterosuperior direction using blunt and sharp techniques until the masseter muscle fibers were exposed.
     6. The facial nerve fibers, though not consistently visible, were preserved and protected during dissection through the deeper layers.
     7. The deeper muscle fibers beneath the facial nerve were transected to provide access to the fracture site.
     8. Once the bone surface was reached, the periosteum was elevated and the fracture identified. Reduction of the fracture segments was facilitated by releasing the IMF and mobilizing the distal segment caudally through intraoral pressure applied to the mandibular molars or by inserting a screw into the ramus and pulling the mandible downwards.
     9. Rigid fixation was achieved by osteosynthesis using 3D-Delta plate:

  <!-- -->

  1. The two superior arm holes of the 3D delta plate were fixed to the proximal segment with two 2.0 mm screws (9mm each) to assist in reduction and manipulation.
  2. The base of the plate was secured to the distal segment with two 2.0 mm screws (7mm each).

     10. Hemostasis was achieved, and the wound was closed in layers. 11. Heavy intermaxillary elastics were applied for three days postoperatively, followed by medium elastics for four days.

     12. In cases of midline deviation, guiding elastics were maintained for an additional week.

     Postoperative Phase

     Postoperative Care and Medications:

     •Amoxicillin with clavulanic acid 1.2 gm and Metronidazole 500 mg, IV, TID for one day.

     • Diclofenac potassium is administered (25 mg -50 mg oral or IV infusion) 1 to 4 times per day.
     * Dexamethasone 4-8mg IV every 8 hours for the first 24 hour .
     * Chlorhexidine mouthwash was prescribed three times daily for 10 days.
     * Oral hygiene instructions were explained to each patient.
     * A liquid and pureed diet was maintained during the period of maxillomandibular fixation (MMF), followed by a soft diet for 4 weeks after MMF removal.
* Follow-up and Postoperative Records:

Radiographic follow-up was performed using computed tomography (CT) scans immediately postoperatively and at three-month intervals.

Clinical follow-up was initiated one week postoperatively, with subsequent evaluations performed at one month and three months postoperatively. At each visit, Pain score, postoperative occlusion, mandibular midline deviation, lateral and protrusive mandibular movements, and maximum opening was assessed. Any unexpected complications were also recorded.

Ethical Considerations:

1. Open reduction and internal fixation of sub condylar fractures is accompanied with complications such as facial nerve injury, parotid gland fistula, permanent scar, infection, pain, edema, and difficulty in mastication following surgical procedure.
2. Risk of Facial injury can be decreased by choosing the appropriate incision and meticulous dissection of the tissues.
3. Parotid gland fistula is avoided by suturing of parotid capsule or by retroparotid retromandibular approach whenever possible.
4. Permanent scar is best minimized by minimal tissue trauma, suturing in layers then the skin will be sutured by Prolene 6-0, Topical antibiotics and topical silicone gel will be prescribed.
5. Post-operative analgesics and anti-inflammatory medications will be given to control pain and edema.
6. Mastication force is enhanced by physiotherapy.
7. Patients are allowed to withdraw from the trial whenever they want to. In this case, they will be surgically managed by conventional plating systems. All patients will be fully informed about the procedures. The risks and benefits will be thoroughly explained to them. No surgery will be performed without written consent.
8. All personal information and data of the patients will be preserved, maintained and stored in a special filing system available in the department. It will not be exposed to anyone that is not included in the surgical team.

The research ethics committee, Faculty of Dentistry Ain Shams University, reviewed the research plan.

ELIGIBILITY:
Inclusion Criteria:

1. Patients at or over 18 years.
2. Unilateral sub condylar fractures. -

Exclusion Criteria:

1. Bilateral sub condylar fractures
2. Pediatric patients.
3. Intracapsular fractures
4. Patients with Uncontrolled systematic conditions. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2024-11-11 (Actual); Primary Completion 2025-07-19 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
posterior vertical height and anatomic reduction using CT | 3 months
  Radiographic evaluation of posterior vertical height and anatomic reduction using CT

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zachariades N, Mezitis M, Mourouzis C, Papadakis D, Spanou A. Fractures of the mandibular condyle: a review of 466 cases. Literature review, reflections on treatment and proposals. J Craniomaxillofac Surg. 2006 Oct;34(7):421-32. doi: 10.1016/j.jcms.2006.07.854. Epub 2006 Oct 19. PMID 17055280
- [Background] Kang DH. Surgical management of a mandible subcondylar fracture. Arch Plast Surg. 2012 Jul;39(4):284-90. doi: 10.5999/aps.2012.39.4.284. Epub 2012 Jul 13. PMID 22872829
- [Background] Ellis E 3rd, Throckmorton G. Facial symmetry after closed and open treatment of fractures of the mandibular condylar process. J Oral Maxillofac Surg. 2000 Jul;58(7):719-28; discussion 729-30. doi: 10.1053/joms.2000.7253. PMID 10883686
- [Background] Tandon S, Verma V, Rashid M, Srivastava S, Singh AK, Sharma NK. Is the facial nerve at risk following surgical correction of mandibular condylar fracture: A systematic review and meta-analysis. Natl J Maxillofac Surg. 2022 Aug;13(Suppl 1):S1-S10. doi: 10.4103/njms.njms_481_21. Epub 2022 Aug 20. PMID 36393942
- [Background] Nys M, Van Cleemput T, Dormaar JT, Politis C. Long-term Complications of Isolated and Combined Condylar Fractures: A Retrospective Study. Craniomaxillofac Trauma Reconstr. 2022 Sep;15(3):246-252. doi: 10.1177/19433875211026759. Epub 2021 Jun 23. PMID 36081681
- [Background] Moloro Michael, Ghali G.E., Larsen PE. Peterson's Principles of Oral and Maxillofacial Surgery . fourth. 2022. 649-670 p
- [Background] Kommers SC, Boffano P, Forouzanfar T. Consensus or controversy? The classification and treatment decision-making by 491 maxillofacial surgeons from around the world in three cases of a unilateral mandibular condyle fracture. J Craniomaxillofac Surg. 2015 Dec;43(10):1952-60. doi: 10.1016/j.jcms.2015.08.031. Epub 2015 Sep 9. PMID 26498515
- [Background] Singh V, Bhagol A, Goel M, Kumar I, Verma A. Outcomes of open versus closed treatment of mandibular subcondylar fractures: a prospective randomized study. J Oral Maxillofac Surg. 2010 Jun;68(6):1304-9. doi: 10.1016/j.joms.2010.01.001. Epub 2010 Apr 3. PMID 20363548
- [Background] Huang CM, Chan MY, Hsu JT, Su KC. Biomechanical analysis of subcondylar fracture fixation using miniplates at different positions and of different lengths. BMC Oral Health. 2021 Oct 21;21(1):543. doi: 10.1186/s12903-021-01905-5. PMID 34674692
- [Background] Ashor M, Salah A, Shindy M, Selim H, Metwaly S, Behairy G. Clinical and radiographic outcomes of rhomboid plate in management of subcondylar fractures: prospective randomized controlled trial. Egypt. J. Oral Maxillofac. surg. 2018 Jan 1;9(1):1-5.
- [Background] Lauer G, Haim D, Proff P, Richter G, Pradel W, Fanghanel J, Pilling E, Gedrange T, Mai R. Plate osteosynthesis of the mandibular condyle. Ann Anat. 2007;189(4):412-7. doi: 10.1016/j.aanat.2007.02.021. PMID 17696004
- [Background] Albogha MH, Mori Y, Takahashi I. Three-dimensional titanium miniplates for fixation of subcondylar mandibular fractures: Comparison of five designs using patient-specific finite element analysis. J Craniomaxillofac Surg. 2018 Mar;46(3):391-397. doi: 10.1016/j.jcms.2017.12.020. Epub 2017 Dec 26. PMID 29311022
- [Background] Chaudhary M, Pant H, Singh M, Vashistha A, Kaur G. Evaluation of trapezoidal-shaped 3-D plates for internal fixation of mandibular subcondylar fractures in adults. J Oral Biol Craniofac Res. 2015 Sep-Dec;5(3):134-9. doi: 10.1016/j.jobcr.2015.07.005. Epub 2015 Aug 15. PMID 26587378
- [Result] Choi KY, Yang JD, Chung HY, Cho BC. Current concepts in the mandibular condyle fracture management part I: overview of condylar fracture. Arch Plast Surg. 2012 Jul;39(4):291-300. doi: 10.5999/aps.2012.39.4.291. Epub 2012 Jul 13. PMID 22872830
- [Result] Ahuja SA, Galinde J, Asnani U, Mistry YA. Comparative Evaluation of Clinical Outcomes Using Delta Plates and Conventional Miniplates for Internal Fixation of Mandibular Condylar Fractures in Adults. J Oral Maxillofac Surg. 2018 Jun;76(6):1255-1266. doi: 10.1016/j.joms.2017.12.018. Epub 2017 Dec 30. PMID 29360455
- [Result] Lata J, Verma N, Mahajan S. Evaluation of Efficacy of 3-Dimensional Delta Versus Trapezoidal Condylar Plates in Internal Fixation of Mandibular Subcondylar Fractures: A Clinical Study. The Traumaxilla. 2019 Apr;1(1):11 21.
- [Result] Sikora M, Sielski M, Stapor A, Chlubek D. Use of the Delta plate for surgical treatment of patients with condylar fractures. J Craniomaxillofac Surg. 2016 Jul;44(7):770-4. doi: 10.1016/j.jcms.2016.04.008. Epub 2016 Apr 15. PMID 27189923
- [Result] Sarkar A, Banerjee L, Ghosh S. Efficacy of Delta Plate in Condylar Fracture: a Case Series with Review. J Dent (Shiraz). 2023 Mar;24(1):71-75. doi: 10.30476/DENTJODS.2022.94746.1806. PMID 36864994

DOCUMENTS (1):
  • Study Protocol: Major issue solved (2023-12-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT07311239/Prot_000.pdf